CLINICAL TRIAL: NCT01037426
Title: Falls and Cardiovascular Events in Elderly Patients With Sinus Node Disease Treated With a MVPTM Pacemaker According to the ESC 2007 Guidelines
Brief Title: Falls and Cardiovascular Events in Pacemaker Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CH190609-V1
Record Dates: First submitted 2009-08-06; First posted 2009-12-23 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-09

CONDITIONS: Bradycardia
Keywords: SND Sinus Node Disease; Falls; Fractures
MeSH Terms: conditions — Bradycardia; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Patients were their own control and number of falls was compared in the year before and after Pacemaker implant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Other): Falls before versus after pacemaker implant
  Interventions: Other: Fill out Questionnaire

INTERVENTIONS:
Other: Fill out Questionnaire — Questionnaire at time of Implantation and 12 months after pacemaker implantation to collect
  * History of falls and fractures during the 12 months before pacemaker implantation
  * Risk markers for falls based on FRAX risk calculator (age, gender, weight, height, history of previous fracture, family history of hip fracture, current smoking habits, glucocorticosteroid intake, rheumatoid arthritis, secondary osteoporosis, alcohol intake)
  * History of falls and fractures during the 12 months after pacemaker implantation
  * Medical and Arrhythmia History
  * Cardiovascular Events
  * Cardiovascular Medication
  * Device programming information

SUMMARY:
The purpose of this study is to document the number of falls and fractures in Sinus Node Disease (SND) patients.

DETAILED DESCRIPTION:
The purpose of this study is to compare the number of falls and fractures in Sinus Node Disease (SND) patients before versus after implantation of a MVP (TradeMark) pacemaker. Further the effect of pacing in the MVP (TradeMark) mode in respect of cardiovascular events is going to be analyzed in the same population.

ELIGIBILITY:
Inclusion Criteria:

* Sinus Node Disease (SND) treated with a pacemaker with MVP (TM) mode according to ESC 2007 guidelines (SND as primary indication for pacemaker implant, implant within past two weeks)
* Geographic stability and availability for follow-up at the study center for the length of the study
* Willingness and Ability to sign Informed Consent

Exclusion Criteria:

* Age less than 50 years
* Impaired cognitive function (such as Alzheimer's disease)
* permanent AV Block II and III
* Persistent atrial fibrillation
* Life expectancy less than two years
* Enrollment or intended participation in another clinical trial during the course of this study
* Subject is pregnant or breastfeeding

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
number of falls in SND patients during one year before versus one year after implantation of a MVPTM pacemaker | 2 years

SECONDARY OUTCOMES:
fracture risk profile and 10-yr fracture risk based on the WHO FRAX index | 2 years
fall rate of recurrent fallers | 2 years
fracture rate | 2 years
combined CV and mortality endpoint | 2 years
any of the individual cardiovascular endpoints | 2 years
mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuehne, Dr. med., Principal Investigator — University Hospital, Basel, Switzerland; Ray Moser, PhD, Study Director — Medtronic (Schweiz) AG - Münchenbuchsee - Switzerland
Locations (8):
- Switzerland (8):
  - Zuger Kantonsspital, Baar
  - University Hospital Basel, Basel
  - SG Spitalregion RWS, Kanton Sankt Gallen
  - Kantonsspital St. Gallen, Sankt Gallen
  - CHCVS - Hôpital de SION, Sion
  - Luzerner Kantonsspital, Sursee
  - Stadtspital Waid, Zurich
  - USZ - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No
there is no plan

REFERENCES:
- [Background] Brenner R, Ammann P, Yoon SI, Christen S, Hellermann J, Girod G, Knaus U, Duru F, Krasniqi N, Ramsay D, Sticherling C, Lippuner K, Kuhne M. Reduction of falls and fractures after permanent pacemaker implantation in elderly patients with sinus node dysfunction. Europace. 2017 Jul 1;19(7):1220-1226. doi: 10.1093/europace/euw156. PMID 27702858